CLINICAL TRIAL: NCT01803438
Title: Catheter Cryoablation Versus Antiarrhythmic Drug as First-Line Therapy of Paroxysmal Atrial Fibrillation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cryo-FIRST
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Symptomatic Paroxysmal Atrial Fibrillation Without Clinically Significant Heart Diseases
Keywords: paroxysmal Atrial Fibrillation; Cryoablation; Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AADs (Active Comparator): AAD therapy based on hospital clinical practice according to ESC Guidelines 2012
  Interventions: Drug: Antiarrhythmic Drugs
- Cryoablation procedure (Experimental): electrical pulmonary veins isolation performed with cryoballoon ablation system
  Interventions: Device: cryoballoon ablation system

INTERVENTIONS:
Device: cryoballoon ablation system
  Arms: Cryoablation procedure
Drug: Antiarrhythmic Drugs — AAD therapy based on hospital clinical practice according to ESC Guidelines 2012
  Arms: AADs

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Pulmonary Vein Isolation (PVI) performed with the Arctic Front™ Advance Cardiac CryoAblation Catheter System as first-line therapy in comparison with antiarrhythmic drugs (AAD) in patients with paroxysmal atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with symptomatic paroxysmal atrial fibrillation as defined above and at least two symptomatic episodes in the last six months prior to inclusion.
* At least one episode of AF must be documented during the prior year by any kind of ECG recording.
* Subject has structural normal heart with an LVEF ≥ 50%, thickness of the inter-ventricular septum ≤12 mm and left atrium diameters (short axis) < 46 mm obtained by transthoracic echocardiography.
* Subject has normal ECG parameters (QRS width in the 12 channel surface ECG ≤120 ms, QTc - interval < 440 ms, PQ - interval ≤ 210 ms; all parameters should be measured at sinus rhythm).
* Subject is at least 18 and not older than 75years old.
* Subject is able and willing to give informed consent.

Exclusion Criteria:

* Subject developed persistent AF at least once in history (electrical or pharmacological cardioversion after 48h or episode duration >7 days).

  * Subject has documented typical atrial flutter.
  * Subject has any history of successful or unsuccessful treatment of AF with class I or III antiarrhythmic or sotalol with the intention to prevent an AF recurrence. Patients pretreated with above AAD at maximum 48 hours with the intention to convert an AF episode are allowed.
  * Subject had any previous left atrial ablation.
  * Subject had any previous cardiac surgery, e.g. prosthetic valves.
  * Subject has permanent pacemaker or defibrillator implant.
  * Subject has 2° type II, 3° degree AV-block or left/right bundle branch block pattern.
  * Subject has unstable angina pectoris.
  * Subject has history of previous myocardial infarction or percutaneous intervention during the last three months.
  * Subject has symptomatic carotid stenosis.
  * Subject has chronic obstructive pulmonary disease with detected pulmonary hypertension or any other evidence of significant lung disease.
  * Subject has any contraindication for oral anticoagulation.
  * Subject has any history of previous transient ischemic attack or stroke.
  * Subject has known intra-cardiac thrombus formation.
  * Subject has any significant congenital heart defect corrected or not (except for patent foramen ovale that is allowed).
  * Subject has evidence of congestive heart failure (NYHA class II, III or IV) in sinus rhythm.
  * Subject has hypertrophic cardiomyopathy.
  * Subject has abnormal long or short QT interval, signs of Brugada syndrome, known inheriting ion channel disease on the family, arrhythmogenic right ventricular dysplasia.
  * Subject has sarcoidosis.
  * Subject has pulmonary vein stent.
  * Subject has myxoma. Exclusion criteria based on laboratory abnormalities
  * Subject has thrombocytosis (platelet count > 600,000 / μl) or thrombocytopenia (platelet count <100,000 / μl).
  * Subject has any untreated or uncontrolled hyperthyroidism or hypothyroidism.
  * Subject has renal dysfunction with glomerular filtration rate < 60 ml / min.
  * Subject has known cryoglobulinaemia. General exclusion criteria
  * Subject has a reversible causes for AF like hyperthyroidism and alcoholism.
  * Subject is a pregnant woman or woman of childbearing potential not on adequate birth control: only woman with a highly effective method of contraception [oral contraception or intra-uterine device] (who must have a negative pregnancy test within 1 week of the start of the therapy) or sterile woman can be enrolled.
  * Subject is a breastfeeding woman.
  * Subject has an active systemic infection.
  * Subject is employed by Medtronic or by the department of any of the investigators or is a close relative of any of the investigators.
  * Subject is unwilling or unable to comply fully with study procedures and follow-up due to any disease condition, which can raise doubt about compliance and influencing the study outcome especially any kind of cancer, severe bleeding in history or a suspected pro-coagulant state.
  * Legal incapacity or evidence that a subject cannot understand the purpose and risks of the study or inability to comply fully with study procedures and follow up.
  * Subject has a life expectancy of ≤ 1 year.
  * Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-06; Primary Completion 2019-10-16 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Freedom from any atrial arrhythmia recurrence | 12 months
  The primary endpoint is freedom from any atrial arrhythmia recurrence at 12 months (at least one episode of AF, atrial flutter or atrial tachycardia with a duration > 30 seconds documented by 7 day Holter ECG or any other printed ECG recording following a blanking period or a dosing optimizing period of 3 months).

SECONDARY OUTCOMES:
quality of life | 12 months
  The quality of life of the two arms measured by means of SF-36 Health Survey and Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) questionnaires will be compared at 12 months follow-up.
Hospital or emergency services accesses | 12 Months
  Hospital or emergency services accesses due to symptoms caused by documented atrial arrhythmias will be compared in the two arms at 12 months follow-up.
Freedom from occurrence of AF | 12 months
  Freedom from occurrence of AF (after 3 months blanking period) will be compared between the two arms at 12 months follow-up.
Freedom from occurrence of documented left atrial tachycardia and left atrial flutter | 12 months
  Freedom from occurrence of documented left atrial tachycardia and typical - or atypical left atrial flutter (after 3 months blanking period or AAD optimization period) will be compared between the two arms at 12 months follow-up.
Symptomatic palpitations burden | 12 months
  Symptomatic palpitations burden will be evaluated by mean of Patient's diary information and compared between the two arms at 12 months follow-up.
Severe adverse events incidence | 12 months
  Severe adverse events incidence will be compared between the two arms during the whole course of the study.
Freedom from persistent AF | 12 months
  Freedom from persistent AF (AF episode lasting longer than 7 days or interrupted by pharmacological or electrical cardioversion after 48h from the onset of the episode) will be compared between the two arms at 12 months follow-up.
Echocardiographic left atrial re-modelling | 12 months
  Echocardiographic left atrial parameters will be compared between the two arms at 6 and 12 months follow ups.
health care utilization | 12 months
  Frequency, type and associated cost of health care utilization and utility will be compared between the two arms at 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kuniss, MD, Principal Investigator — Kerckhoff - Klinik, Bad Nauheim, Germany; GianBattista Chierchia, MD, Principal Investigator — Heart Rhythm Management Centre, UZ Brussels - VUB Brussel, Belgium
Locations (19):
- nstituto Cardiovascular de Buenos Aires, Buenos Aires, Argentina
- Monash Medical Centre, Melbourne, Australia
- Heart Rhythm Management Centre, UZ Brussels - VUB Brussel, Brussels, Belgium
- Croatia (2):
  - Klinicki bolnicki centar Sestre Milosrdnice, Zagreb
  - Klinicki bolnicki centar Sestre, Zagreb
- France (4):
  - NCHU Amiens, Amiens
  - CHU Grenoble, Grenoble
  - CHU La Pitié, Paris
  - CHU Charles Nicolle, Rouen
- Germany (5):
  - Kerckhoff - Klinik, Bad Nauheim
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Universitätsklinikum Eppendorf, Hamburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Klinikum Bogenhausen, Munich
- Italy (2):
  - Maria Cecilia Hospital, Cotignola
  - Ospedale S.S. Giacomo e Cristoforo, Massa
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus MC, Rotterdam
- Haukeland Hospital, Bergen, Norway

REFERENCES:
- [Derived] Andrade JG, Moss JWE, Kuniss M, Sadri H, Wazni O, Sale A, Ismyrloglou E, Chierchia GB, Kaplon R, Mealing S, Bainbridge J, Bromilow T, Lane E, Khaykin Y. The Cost-Effectiveness of First-Line Cryoablation vs First-Line Antiarrhythmic Drugs in Canadian Patients With Paroxysmal Atrial Fibrillation. Can J Cardiol. 2024 Apr;40(4):576-584. doi: 10.1016/j.cjca.2023.11.019. Epub 2023 Nov 23. PMID 38007219
- [Derived] Pavlovic N, Chierchia GB, Velagic V, Hermida JS, Healey S, Arena G, Badenco N, Meyer C, Chen J, Iacopino S, Anselme F, Dekker L, Scazzuso F, Packer DL, de Asmundis C, Pitschner HF, Piazza FD, Kaplon RE, Kuniss M; Cryo-FIRST Investigators. Initial rhythm control with cryoballoon ablation vs drug therapy: Impact on quality of life and symptoms. Am Heart J. 2021 Dec;242:103-114. doi: 10.1016/j.ahj.2021.08.007. Epub 2021 Sep 8. PMID 34508694